CLINICAL TRIAL: NCT00575328
Title: A Double-Blind, Placebo Controlled Study of Maca Root for the Treatment of Sexual Dysfunction Associated With the Treatment Regimen for Bipolar Disorder in Females
Brief Title: Study of Maca Root to Treat Sexual Dysfunction Associated With the Treatment Regimen for Bipolar Disorder in Females
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Only N=8 subjects randomized; funding ran out; too small N to yield useful data.
Sponsor: Massachusetts General Hospital (Other)
Collaborators: National Alliance for Research on Schizophrenia and Depression (Other)
Responsible Party: Principal Investigator, David Mischoulon, MD, PhD, MD, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2007-P-001471
Record Dates: First submitted 2007-12-14; First posted 2007-12-18 (Estimated); Results first posted 2020-09-07 (Actual); Last update posted 2020-09-25 (Actual); Status verified 2020-09

CONDITIONS: Sexual Dysfunction; Bipolar Disorder
Keywords: Sexual Dysfunction; Bipolar Disorder
MeSH Terms: conditions — Sexual Dysfunction, Physiological; Bipolar Disorder

STUDY DESIGN:
Intervention Model Description: Maca root will be compared against inactive placebo as a treatment for sexual dysfunction induced by psychotropic drugs.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: All subjects, investigators, and clinical assessors were blinded to the intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Maca Root (Experimental): Subjects in this arm will be given 3g/day of Maca Root.
  Interventions: Drug: Maca Root
- Placebo (Placebo Comparator): Subjects in this arm will receive inactive placebo.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Maca Root — 3g/day of Maca Root for 12 weeks.
  Other Names: Lepidium
  Arms: Maca Root
Drug: Placebo — Placebo provided by research pharmacy daily for 12 weeks.
  Other Names: Inactive placebo
  Arms: Placebo

SUMMARY:
The purpose of this research study is to find out whether Maca Root is effective for treating sexual dysfunction in females that is caused by the treatment for bipolar disorder. An additional aim of the study is to document the safety and tolerability of maca root, as well as any potential side effects that it causes. We suspect that Maca Root will result in a significant reduction in sexual dysfunction when compared to a placebo group.

DETAILED DESCRIPTION:
The study seeks to enroll 80 patients with sexual dysfunction associated with their bipolar medication regimen over 24 months. Subjects were outpatient females between 18 and 80 years old with no significant symptoms of mania (Young Mania Rating Scale score<10), and who have been on a steady regimen of medications to treat bipolar disorder for at least 8 weeks, with a stable dose for at least 4 weeks. Subjects will be randomly assigned in a double blind manner to receive 3000 mg/day of maca root or identical placebo for 12 weeks to determine whether maca root is more effective than placebo for the treatment of sexual dysfunction associated with treatment regimens for bipolar disorder.

ELIGIBILITY:
Inclusion Criteria:

* Subject is female, age 18 to 80 years
* Subject has been on a steady regimen to treat bipolar disorder, including monotherapy with or any combination of antidepressants, mood stabilizers, atypical antipsychotics, or benzodiazepines, for at least 8 weeks; and is currently on a stable dose of that regimen for at least 4 weeks
* Subject is currently euthymic (Hamilton-D scale score < 10) and is without significant anxiety symptoms (Hamilton-A < 10). Her bipolar disorder must be in remission (Young Mania Rating Scale score < 10)
* Subject must have had no sexual dysfunction prior to taking psychotropic medications and there must be a clear temporal relationship between the sexual dysfunction and the treatment for bipolar disorder
* Subject must have been consistently experiencing at least one of the following criteria for at least 4 weeks, with distress or disability:
* Inability to have an orgasm, according to patient opinion
* Clinically significant orgasm delay with masturbation or intercourse
* Inability to attain or maintain until completion of sexual activity an adequate lubrication swelling response of sexual excitement
* Decreased libido according to patient opinion
* Subject must be having or had been having some form of regular sexual activity (masturbation, oral sex, intercourse) at least twice monthly prior to the bipolar treatment regimen and is willing to continue efforts at sexual activity at least once weekly for the duration of the study
* Subject must be in good general physical health
* Subject must be able to understand and communicate in English
* Subject must have given informed consent to participate in the study

Exclusion Criteria:

* Primary or prior diagnosis of a sexual disorder (other than the side effect of the bipolar medication or symptom of the bipolar disorder)
* Sexual dysfunction secondary to general underlying medical condition
* Penile, vaginal, clitoral or other sexual organ anatomical deformities
* Any uncontrolled psychiatric disorder
* Alcohol or substance abuse or dependence within the past six months
* Recent major relationship changes, disruption, or turmoil ongoing or anticipated which are unrelated to her sexual dysfunction
* Blood pressure outside the range of 90/50 - 170/100
* Known hyperprolactinemia
* Use of investigational drugs within previous 3 months or during study
* Current use of other drugs for sexual dysfunction or other therapies or medications to treat sexual dysfunction
* Current use of nefazodone
* Hormone replacement therapy, unless patient has been on stable dose of hormone therapy for at least 3 mo prior to the bipolar treatment regimen and had no sexual dysfunction while on the same hormone therapy regimen, and there is no change in the hormone replacement therapy during the study
* Pregnancy, lactating, or planning to become pregnant during the study
* Child bearing potential subjects unwilling and/or not prepared and/or who are judged unreliable to use an acceptable and verifiable form of contraception during the study
* Any clinically significant abnormality on the screening physical examination
* History of hormonal cancers
* Any medical or psychological condition or social circumstances that would impair subject's ability to participate reliably in the study, or that may increase the risk to subjects or others as a result of participating in this study
* Dyspareunia secondary to an inflammatory or anatomical condition
* Prior use of maca for at least two weeks
* Infection of the urogenital tract that may make sexual activity painful or difficult
* Subjects whose sexual partners are suffering from and/or receiving treatment for sexual dysfunction
* Receiving psychosexual or other therapy for sexual dysfunction and not willing to discontinue that treatment at screening
* Subjects who do not understand and communicate in English
* Subjects for whom sexual activity is inadvisable
* Subjects whose sexual dysfunction is considered to be situational
* Subjects not attempting some form of regular sexual activity at least twice monthly and at least once weekly during study visit intervals for duration of entire study
* Changes in bipolar medication and/or dose of medication within the last 4 weeks before baseline visit
* Participants on medications with a narrow therapeutic window or low therapeutic index for which small variations may be harmful given the lack of systematic experience with drug-supplement interactions (i.e. - cyclosporine, digoxin, warfarin, and antiretrovirals)

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2008-02-26 (Actual); Primary Completion 2010-04-26 (Actual); Study Completion 2010-04-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christina Dording, MD, Principal Investigator — Massachusetts General Hospital; David Mischoulon, MD, PhD, Study Director — Massachusetts General Hospital
Locations (1):
- Depression Clinical and Research Program, Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No
No plan for data sharing at this time. Study was never completed and did not have enough subjects to yield useful data.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Female subjects with remitted bipolar disorder and sexual dysfunction associated with their bipolar medication treatment regimens were recruited from 2/26/2008 to 4/26/2010, all at the Massachusetts General Hospital Depression Clinical and Research Program.
Pre-assignment Details: Subjects underwent a screening visit to determine eligibility. Those subjects deemed eligible returned a week later for a baseline visit, where eligibility was confirmed prior to treatment assignment. Subjects who for any reason no longer met entry criteria were discontinued and offered alternative treatment options.
Period: Overall Study
Arm/Group | Maca Root | Placebo
Started | 4 | 4
Completed | 1 | 2
Not Completed | 3 | 2
Not completed — Adverse Event | 1 | 1
Not completed — Lost to Follow-up | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Maca Root | Placebo | Total
Number analyzed (Participants) | 4 | 4 | 8
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 4 | 4 | 8
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 37 (11) | 37 (10) | 37 (10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 4 | 8
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 4 | 3 | 7
  Asian-Hispanic | 0 | 1 | 1
Region of Enrollment [Count of Participants; unit: Participants] — Location: Massachusetts General Hospital, Depression Clinical and Research Program, Boston, Massachusetts, USA
  Participants
    United States | 4 | 4 | 8
Hamilton D-17 score [Mean (Standard Deviation); unit: units on a scale] — The 17-item Hamilton Rating Scale for Depression (HAM-D-17) is a structured interview completed by the clinician based on assessment of patient's depressive symptoms. It quantifies degree and severity of depression. Higher scores indicate greater pathology. Possible range of scores is from zero (no symptoms) to 52 (very severe symptoms). Scores of 10 or less are considered to have no significant depression (11-15=mild, 16-22=moderate, >23= severe). For entry, subjects were required to have a score of less than 10.
  units on a scale | 6 (3) | 6 (2) | 6 (2)
Young Mania Rating Scale score [Mean (Standard Deviation); unit: units on a scale] — Young Mania Rating Scale (YMRS) has 11 items to assess severity of mania in patients with bipolar disorder. The items in this scale reflect core symptoms of the manic phase of bipolar disorder. YMRS total score ranges from 0 to 60; higher scores indicate more severe mania, thus, a negative change (or decrease) from baseline indicates a reduction in manic symptoms. Total score ≤12 indicates remission (13-19=minimal symptoms; 20-25=mild mania, 26-37=moderate mania, 38-60=severe mania). Scores <10 are considered fully euthymic. For entry, subjects were required to have a score of less than 10.
  units on a scale | 2 (1.8) | 1.5 (1.7) | 1.8 (1.7)

OUTCOME MEASURES:

1. Primary Outcome: Reductions in Arizona Sexual Experience Scale (ASEX) Scores Over 12 Weeks of Treatment.
Description: The ASEX scale consists of five items rating sexual drive, arousal, vaginal lubrication/penile erection, ability to reach orgasm, and satisfaction from orgasm. The range of total score is from 5-30, with the higher scores indicating greater sexual dysfunction. Scores were obtained at baseline and at all biweekly assessment visits over the 12 weeks of treatment.
Time Frame: Biweekly from Baseline (week zero) to 12 weeks
Population: Intent to treat sample. Subjects with at least one post baseline visit recorded with available data.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Maca Root | Placebo
Number analyzed (Participants) | 3 | 3
units on a scale
  ASEX-Baseline Score | 23.7 (1.5) | 21.3 (0.6)
  ASEX-Final Score | 23.3 (3.8) | 23 (2.8)
  ASEX-Change in Score | -0.3 (4.2) | 1.5 (2.1)
Statistical Analysis 1: Comparison: Maca Root vs Placebo; Null hypothesis: There will be no difference in clinical improvement (i.e. change in ASEX score) between treatment arms. No formal power analysis was carried out, given the small study sample; Test type: Superiority — Analysis is a test of statistical significance to evaluate whether the results are consistent with the assumption of there being no difference in the clinical improvement (i.e. change in ASEX score) of the two treatments (null hypothesis); p = 0.62, t-test, 2 sided — No adjustment for multiple comparisons. P value for significance set a priori at P<0.05; Mean Difference (Final Values) = 1.8, 95% CI 2-sided [-8.7 to 12.3], Standard Deviation 3.3; The analysis is not truly informative, since the analyzable sample (n=6) was too small. Results should be viewed with caution

2. Primary Outcome: Reductions in Massachusetts General Hospital Sexual Dysfunction (MGH-SD) Inventory Scores Over 12 Weeks of Treatment.
Description: This instrument is composed of five items evaluating libido, sexual arousal or excitement, ability to achieve orgasm, ability to achieve and maintain an erection (for men only) and overall sexual satisfaction. Items are rated on a scale of 1 to 6 with a rating of 1 indicating greater than normal functioning and a rating of 6 indicating totally absent functioning. Possible total scores range from 5-30, with higher scores indicating greater pathology. Scores were obtained at baseline and at each biweekly assessment visit over 12 weeks of treatment.
Time Frame: Biweekly from Baseline (week zero) to 12 weeks
Population: Intent to treat sample. Subjects with at least one post baseline visit recorded with available data.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Maca Root | Placebo
Number analyzed (Participants) | 3 | 3
units on a scale
  MGH-SD Score-Baseline | 21 (2) | 18.7 (2.3)
  MGH-SD Score-Final | 16.7 (5.0) | 18 (1.7)
  Change in MGH-SD Score | -4.3 (6.1) | -0.7 (2.1)
Statistical Analysis 1: Comparison: Maca Root vs Placebo; Null hypothesis: There will be no difference in clinical improvement (i.e. change in MGH-SD score) between treatment arms. No formal power analysis was carried out, given the small study sample; Test type: Superiority — Analysis is a test of statistical significance to evaluate whether the results are consistent with the assumption of there being no difference in the clinical improvement (i.e. change in MGH-SD score) of the two treatments (null hypothesis); p = 0.38, t-test, 2 sided — No adjustment for multiple comparisons. P value for significance set a priori at P<0.05; Mean Difference (Final Values) = 3.6, 95% CI 2-sided [-6.7 to 13.97], Standard Deviation 4.5; Analysis was not truly informative since the analyzable sample (n=6) was too small. Results should be interpreted with caution

ADVERSE EVENTS:
Time Frame: 2 years.
Description: All adverse events were systematically recorded and reported to the Institutional Review Board (IRB). All significant adverse effects were immediately reported upon their discovery and monitored through the following methods: 1) Going over any adverse events with the patient at each study visit 2) holding weekly meetings with the principal investigator and study staff team to review all safety and tolerability issues that were brought up.
Arm/Group | Maca Root | Placebo
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/4
Serious Adverse Events (participants affected / at risk) | 1/4 | 0/4
Other Adverse Events (participants affected / at risk) | 3/4 | 2/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Maca Root (N=4) | Placebo (N=4)
Menorrhagia (Reproductive system and breast disorders) | 1 (1) | 0 (0) — Severe bleeding during menstrual period.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Maca Root (N=4) | Placebo (N=4)
Bloating (Gastrointestinal disorders) | 0 (0) | 1 (1) — Sensation of bloating
Heartburn symptom (Gastrointestinal disorders) | 0 (0) | 2 (2) — General stomach upset
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) — Nausea sensation
Vaginal bleeding (Reproductive system and breast disorders) | 0 (0) | 2 (2) — Mild bleeding from vagina outside of regular menstrual periods.
Influenza (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) — Flu
Upper Respiratory Infection (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) — Common cold
Sore throat (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) — Sore throat in absence of other upper respiratory symptoms.
Fatigue (General disorders) | 1 (1) | 0 (0) — Generalized fatigue
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0) — increased generalized anxiety
Forgetfulness (Nervous system disorders) | 1 (1) | 0 (0) — Generalized forgetfulness of tasks, appointments.
Superficial laceration of leg (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) — Accidental cut on leg

LIMITATIONS AND CAVEATS:
Study was never completed due to low enrollment. Only 8 of a projected 80 subjects were randomized over a period of 2 years. Sample is too small to yield useful information.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No